CLINICAL TRIAL: NCT06811948
Title: Sleep-Disordered Breathing in the Acute Phase After Stroke and Neuropsychiatric Outcomes
Status: Not yet recruiting | Type: Observational
Sponsor: Blekinge County Council Hospital (Other)
Responsible Party: Principal Investigator, Joseph Aked, Post-doc, Resident Physician Internal Medicine, Blekinge County Council Hospital
Other Study IDs: 2024-02659-01
Record Dates: First submitted 2025-01-27; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Stroke; Fatigue Symptom; Obstructive Sleep Apnea; Sleep Disordered Breathing (SDB)
MeSH Terms: conditions — Stroke; Fatigue; Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In people who have had a stroke or a transient ischemic attack (TIA), it is common to have problems with breathing patterns during sleep, particularly a condition called obstructive sleep apnea. Another common long-term problem after a stroke is post-stroke fatigue, which affects function and quality of life after stroke. There is currently no clearly effective treatment for post-stroke fatigue. We are investigating whether there might be a connection between sleep-related breathing disturbances, and the risk of developing long-term post-stroke fatigue

The project is being conducted at Blekingesjukhuset Karlskrona, and inpatients with stroke are asked to participate. Participants are equipped with a sleep analysis pad under the mattress that measures breathing patterns during the night, as well as a wrist-worn device that measures oxygen saturation in the blood. Participants are also asked about their functional level in daily life and any symptoms of obstructive sleep apnea. One year after the stroke, participants are invited for a follow-up visit where we ask about post-stroke fatigue, depressive symptoms, and treatment and investigations related to the stroke.

We will then investigate the relationship between sleep-related breathing disturbances, measured early after stroke, and the risk of significant fatigue after the stroke. This could lead to future studies with treatment trials for obstructive sleep apnea in certain individuals with post-stroke fatigue. The study could also lead to potentially increased awareness that these conditions might be connected, which could result in a higher likelihood of detecting treatable obstructive sleep apnea in certain subgroups after stroke.

DETAILED DESCRIPTION:
Stroke is the second leading cause of death and a common cause of acquired disability worldwide, and the burden of the disease at the societal level is expected to increase in the coming decades. Stroke can result in various long-term consequences, both neurological (such as aphasia, paresis, sensory or visual disturbances, and coordination and balance disorders) and neuropsychiatric (such as cognitive impairment, depression, and fatigue). These consequences, in turn, affect stroke survivors' physical functions, activity levels, and ability to participate in daily activities.

Post-stroke fatigue is common, with prevalence estimates ranging between 25-85%, and 40% of stroke survivors have reported it as one of their worst symptoms. Recent Swedish studies have estimated the long-term prevalence 3-5 years after stroke to be between 24-52%. Post-stroke fatigue partially overlaps with post-stroke depression, but approximately 70% of individuals with significant fatigue do not exhibit concurrent depressive symptoms . The condition is associated with poorer performance in daily activities and lower health-related quality of life. Currently, there are no specific treatments for post-stroke fatigue. Due to its high prevalence and consequences, it has recently been identified as one of the top ten priority research questions in stroke rehabilitation by the UK National Institute for Health and Care Research.

There are conflicting reports on whether traditional vascular risk factors such as hypertension, hyperlipidemia, heart disease (including atrial fibrillation), and smoking contribute to post-stroke fatigue. Obesity is associated with post-stroke fatigue, and sleep-disordered breathing (SDB) has also emerged as a potential risk factor.

Sleep-disordered breathing is prevalent after stroke, occurring in 50-70% of some populations. The dominant condition is obstructive sleep apnea syndrome (OSAS), followed by central sleep apnea. Established treatments for OSAS include continuous positive airway pressure (CPAP), mandibular advancement devices, surgical interventions, and weight loss, which can reduce daytime sleepiness. Research is ongoing regarding the extent to which treated OSAS can contribute to secondary prevention in stroke. Current American guidelines for secondary prevention provide a class 2b recommendation with moderate evidence for considering OSAS screening after stroke or transient ischemic attack (TIA).

The diagnosis is primarily made through overnight respiratory monitoring, with polysomnography being the gold standard, although it is time- and resource-intensive and may be cumbersome for the patient. Limited polygraphic examinations can also be conducted both in hospitals and at home.

Research Questions:

1. What is the 1-year prevalence of post-stroke fatigue in a hospital-based cohort in Blekinge?
2. How many individuals with stroke have significant sleep-disordered breathing according to non-invasive measurement?
3. What proportion of individuals with post-stroke fatigue had significant sleep-disordered breathing during hospitalization?
4. Can early, non-invasive, and simple measurement of sleep-disordered breathing in hospitals predict a subgroup of stroke patients who will develop significant fatigue?
5. Is there evidence that treatment goals after stroke are achieved to a lesser extent in those with significant fatigue?

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Stroke according to WHO definition (31) (ischemic stroke, intracerebral hemorrhage, or subarachnoid hemorrhage)
* TIA with MRI-verified lesions corresponding to symptoms
* Informed consent to participate

Exclusion Criteria:

* Traumatic stroke
* Tumor-associated bleeding
* Expected survival <3 months
* Unconsciousness (RLS >3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital-based, prospective inclusion at a single site in Karlskrona, Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2027-05-20 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
Fatigue Assessment Scale | 1 year follow-up
  Measurement of post-stroke fatigue at 1 year follow-up.

OTHER OUTCOMES:
Apnea-hypopnea index | Within 72 hours of ictus
  Apnea-hypopnea index measured during hospital stay with Withings Sleep Analyzer. Used as a biomarker for sleep disordered-breathing.
Nocturnal time under 90% blood oxygen saturation | Within 72 hours of ictus
  Measured with pulse oximeter. Used as a biomarker of sleep-disordered breathing.
Oxygen Desaturation Index | Within 72 hours of ictus
  Measure of nocturnal desaturations

CONTACTS AND LOCATIONS:
Locations (1):
- Blekinge Hospital, Karlskrona, Blekinge County, Sweden

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-01-31): https://cdn.clinicaltrials.gov/large-docs/48/NCT06811948/Prot_000.pdf